CLINICAL TRIAL: NCT06064591
Title: Host Immune and Metabolic Determinants of Sexual Conversion in Plasmodium Parasites IMMETASEX
Acronym: IMMETASEX
Status: Recruiting | Type: Observational
Sponsor: Institute of Tropical Medicine, Belgium (Other)
Collaborators: Instituto Nacional de Saúde, Mozambique (Other Government); Clinical Research Unit of Nanoro (CRUN), Burkina Faso (Unknown); Barcelona Institute for Global Health (Other); Leiden University Medical Center (Other); KU Leuven (Other)
Responsible Party: Sponsor
Other Study IDs: IMMETASEX 1704/23; G067823N (Other Grant/Funding Number: FWO Belgium)
Record Dates: First submitted 2023-09-26; First posted 2023-10-03 (Actual); Last update posted 2024-02-01 (Actual); Status verified 2024-01

CONDITIONS: Severe Malaria; Uncomplicated Malaria; Asyptomatic Plasmodium Infection
MeSH Terms: conditions — Malaria

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Days
Biospecimen Retention: Samples With DNA — Venous blood sample
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (7):
- Pilot study Belgium Patients: Patients (P. falciparum-infected)
  No intervention 6 ml of venous blood sampled at one time point
- Pilot study Belgium Controls: Control non-infected individuals No intervention 6 ml of venous blood sampled at one time point
- Work package 1 Burkina Faso Asymptomatic: Asymptomatic (P. falciparum-infected) No intervention Venous blood sample (maximum of 8 ml) at 1 time point. 300µl of finger prick blood at four follow-up visits 24, and 48 and 72h and day 10 after the enrollment.
- Work package 1 Burkina Faso uncomplicated patients: uncomplicated patients (P. falciparum-infected) No intervention Venous blood sample (maximum of 8 ml) at 1 time point.
- Work package 1 Burkina Faso Controls: Control non-infected individuals No intervention Venous blood sample (maximum of 8 ml) at 1 time point.
- Work package 2 Mozambique Uncomplicated malaria patients: Uncomplicated malaria patients No intervention Venous blood sample (maximum of 6 ml) at 1 time point.
- Work package 2 Mozambique Severe malaria patients: Severe malaria patients No intervention Venous blood sample (maximum of 6 ml) at 1 time point.

SUMMARY:
Understanding the sexual conversion of the malaria parasite is essential to interrupt malaria transmission. A new tool is developed that, based on expression analysis of sexual stage biomarkers, will estimate sexual conversion rates in natural infections.

DETAILED DESCRIPTION:
Understanding the sexual conversion of the malaria parasite is essential to interrupt malaria transmission. At each replicating cycle within erythrocytes, a proportion of asexual parasites converts into non-replicative sexual stages, which are the only forms able to infect mosquitos. The rate at which sexual stages are produced, is known as basal sexual conversion rate. Changes in the host immune and metabolic environment associated with the development of malaria disease, such as depletion of lysophosphatidylcholine in plasma, have been associated with increased sexual conversion rates in vitro. It is hypothesised that immune and metabolite factors that are altered during malaria infection induce sexual conversion in Plasmodium falciparum parasites. In this project, a new tool is developed that, based on expression analysis of sexual stage biomarkers, will estimate sexual conversion rates in natural infections. The aim is to identify immune factors and metabolites that induce sexual conversion using in-house developed sexual conversion assays, and experimental mosquito infections. Finally, transcriptional mechanisms are explored driving parasite sexual conversion in the host environment during disease using single-cell RNA-sequencing approaches. This research will provide essential knowledge on the factors that affect sexual conversion in the host and potentially inform novel strategies to interrupt transmission.

ELIGIBILITY:
Inclusion Criteria:

* Age: ≥ 1 year
* Willing and able to provide written informed consent (or assent for minors with written informed consent by parent(s) and/or guardian(s).

Pilot:

-symptomatic for P. falciparum

-/Travel to P. falciparum endemic area within the last month

WP1:

* Resident in Nanoro district
* non-symptomatic individuals

WP2:

* Positive for P. falciparum infection via Rapid Diagnostic Tests (RDT)
* Age: ≥ 1 and ≤ 12 years
* Patients are included when suspected of the following conditions:

I. Severe malaria by infection with P. falciparum is defined in the presence of P. falciparum asexual parasitemia, and as one or more of the following:

1. Impaired consciousness: A Blantyre coma score < 3 (when patients are ≤ 6 years) or Glasgow coma score < 10 (when patients are ≥ 6 years).
2. Prostration: Generalized weakness so that the person is unable to sit, stand or walk without assistance.
3. Multiple convulsions: More than two episodes within 24 hours.
4. Clinical manifestation of respiratory distress (e.g., rapid, deep and labored breathing).
5. Diagnosis through exclusion: absence of an identified alternative cause.

II. Uncomplicated malaria by infection with P. falciparum is defined as a patient who presents with lethargic profile (e.g. fever) and a positive parasitological test for P. falciparum, but with no features of severe malaria.

Exclusion Criteria:

* Delayed developmental status or history of chronic illness
* Participation in another study
* Previous malaria treatment or prophylaxis in the last week
* Inability or unwillingness of the parents or guardians to provide informed consent

WP1:

* Symptoms of malaria, as defined by presence of fever (body temperature >37.5 °C or history of fever during the past 48 hours) with a positive RDT (RDT are performed always when there is presence of fever)
* Any plans to leave the study are in the coming 10 days

WP2:

* Severe anemia (will be determined via clinical examination), since blood samples can hardly be withdrawn, co-morbidities.
* A questionnaire will be used during the clinical assessment that addresses following exclusion criteria:

x Antimalarial drug treatment or other medication during the past week x If the patient had a meal within 4 hours before admission x Patients with acute meningitis (as clinically evaluated according to the local guidelines) x Patients with developmental delay or history of chronic illness x Vaccination during the past week

Min Age: 1 Year | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Pilot:
  This study will be performed at the policlinic of ITM, in Antwerp, Belgium.
  WP1 Recruitment screenings will be organized in Nanoro village, within the catchment area of the existing health demographic surveillance system (HDSS) of Nanoro Health district (NHD), Burkina Faso.
  WP2 The study will include pediatric patients with uncomplicated and severe malaria (aged ≥ 1 and ≤ 12 years, male and female) visiting Chókwè Rural Hospital, Mozambique, and the peripheral health centers in Chókwè district.
Sampling Method: Non-Probability Sample
Enrollment: 430 (Estimated)
Dates: Start 2023-12-13 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
To validate a Sexual Conversion Estimator tool | 2023-2025
  To validate a Sexual Conversion Estimator tool to accurately estimate SC rates and future transmission potential in epidemiological samples. First, the investigators will measure expression levels of SRBs and directly determine SC rates in samples from malaria asymptomatic patients. Second, the investigators will use a machine learning classifier to determine the combination of SRBs that best predicts SC rates; and third, the investigators will measure the predictive value of the Estimator tool for future transmission potential

SECONDARY OUTCOMES:
To investigate in malaria patients associations between host immune and metabolic factors and P. falciparum sexual conversion and infection potential | 2023-2025
  In patients with uncomplicated and severe malaria, the investigators will investigate associations between host inflammatory molecules, parasite-specific Ab and metabolic factors, with parasite SC rates. The investigators hypothesize that SC rates will be higher in severe malaria patients and associated with specific molecules and metabolites.
To validate associations between sexual conversion and host immune and metabolic factors in vitro | 2024-2026
  An in vitro assay, based on recently described gametocyte-reporter parasite lines 16 will be used to validate candidate associations identified in Objective 2. First, the effect of patient serum samples and specific metabolites and inflammatory factors via in vitro SC assays is tested. Next, in vitro cultures with significantly induced SC will be fed to Anopheles stephensi mosquitoes to assess infection potential via standard membrane feeding assays. It is hypothesized that plasma/factors identified in Objective 2, induce SC in vitro and increase mosquito infections.
To explore transcriptional mechanisms driving parasite sexual conversion in the host environment during uncomplicated and severe malaria disease | 2024-2026
  Use of a single cell RNA-sequencing (scRNA-seq) approaches to generate the first in-depth characterization of gene expression patterns of very early sexual stages in the host circulation during natural infections in uncomplicated and severe clinical presentations (samples collected in Objective 2).

CONTACTS AND LOCATIONS:
Overall Officials: Anna Rosanas-Urgell, Prof, Principal Investigator — ITM
Locations (3):
- Institute of Tropical Medicine Antwerp, Antwerp, Belgium
- Institut de Recherche en Sciences de la Santé - Clinical Research Unit of Nanoro, Nanoro, Burkina Faso
- Instituto Nacional de Saúde (INS), Maputo, Mozambique